CLINICAL TRIAL: NCT00303654
Title: Quality Assessment of the Roei Loop Resectoscope for Transurethral Resection of Bladder Neoplasm and BPH
Brief Title: Loop Resectoscope in Treating Patients With Bladder Cancer or Benign Prostatic Hyperplasia Who Are Undergoing Transurethral Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roei Medical Technologies Ltd. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000446284; UCLA-0506127-01
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2007-06

CONDITIONS: Bladder Cancer
Keywords: recurrent bladder cancer; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Biopsy

INTERVENTIONS:
Procedure: biopsy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Transurethral resection is a less invasive type of surgery for bladder cancer or benign prostatic hyperplasia. Transurethral resection using a loop resectoscope may have fewer side effects and improve recovery.

PURPOSE: This clinical trial is studying how well the loop resectoscope works in treating patients with bladder cancer or benign prostatic hyperplasia who are undergoing transurethral resection.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy, in terms of mechanical capabilities, of the Roei loop resectoscope in patients with bladder cancer or benign prostatic hyperplasia undergoing transurethral resection of bladder tumor or benign prostatic adenoma.
* Determine the quality of specimens submitted for histological analysis from patients undergoing this procedure.

OUTLINE: This is an open-label, pilot study.

Patients undergo transurethral resection using the Roei loop resectoscope. Surgeon satisfaction with the Roei loop resectoscope is measured by a self-assessment questionnaire. The quality of specimens submitted for histological study are also assessed.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of bladder cancer or benign prostatic hyperplasia

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-08; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Surgeon satisfaction with usage of Roei loop resectoscope measured by a questionnaire after the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Allan Pantuck, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States